CLINICAL TRIAL: NCT06845072
Title: Validity and Reliability a Low-cost Handgrip Dynamometer in Healthy Adults
Brief Title: Low-Cost Handgrip Dynamometer in Healthy Adults
Status: Active, not recruiting | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Pelin Tiryaki, Physical Therapist, University of Yalova
Other Study IDs: 2024/293
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Hand Grip Strength
Keywords: dynamometer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The gold standard device for measuring grip strength is the Jamar® Hydraulic Hand Dynamometer. The Jamar® Hydraulic Hand Dynamometer is a high-priced device. It has an analog reading feature. The Jamar hydraulic hand dynamometer is recommended by the American Association of Hand Therapists and is considered the gold standard because of its high validity and reliability. Due to its cost, the use of this dynamometer is quite limited in certain countries and settings. However, there is a new version, the JAMAR Plus+, which has a digital reading feature. This version is even more expensive. In recent years, the use of less expensive dynamometers for measuring grip strength has become increasingly common in clinical settings and scientific research. In particular, the Camry Dynamometer, which is ten times cheaper, is frequently used. Despite its frequent use in scientific research, a review of the current literature has shown that the validity and reliability of the Camry has not been examined in healthy populations. Our study compares the Jamar® Hydraulic Hand Dynamometer, the gold standard device for measuring grip strength, with the lower cost and lighter handheld digital Camry dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Healty volunteers with 18-65 years

Exclusion Criteria:

* Using any assistive device,
* Having rheumatoid arthritis, gout, neuromuscular disease or any acute/chronic disease that may affect grip strength,
* Pregnancy,
* Previous subluxation, dislocation or fracture in the upper extremity,
* Type 1 or Type 2 DM,
* Unstable chronic and systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Maximum handgrip strength - Device 1 | 7 days
  Maximum grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles.
Maximum handgrip strength - Device 2 | 7 days
  Maximum grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | Baseline
  The purpose of the questionnaire is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity. The total score is grouped as inactive (<600 MET-min/week), minimally active (minimum 600 MET-min/week and <3000 MET-min/week) and active (>3000 MET-min/week).
SBQ - Sedentary Behaviour Questionnaire | Baseline
  The SBQ was designed to assess the amount of time spent doing 9 behaviors (watching television, playing computer/video games, sitting while listening to music, sitting and talking on the phone, doing paperwork or office work, sitting and reading, playing a musical instrument, doing arts and crafts, sitting and driving/riding in a car, bus, or train). The 9 items were completed separately for weekdays and weekend days.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Tiryaki, PhD, Principal Investigator — University of Yalova
Locations (2):
- Turkey (Türkiye) (2):
  - University of Yalova, Yalova
  - Yalova University, Yalova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cildan Uysal S, Tonak HA, Kitis A. Validity, reliability and test-retest study of Grip strength measurement in two positions with two dynamometers: Jamar(R) Plus and K-Force(R) Grip. Hand Surg Rehabil. 2022 Jun;41(3):305-310. doi: 10.1016/j.hansur.2022.02.007. Epub 2022 Mar 10. PMID 35283336
- [Background] Guerra RS, Amaral TF, Sousa AS, Fonseca I, Pichel F, Restivo MT. Comparison of Jamar and Bodygrip Dynamometers for Handgrip Strength Measurement. J Strength Cond Res. 2017 Jul;31(7):1931-1940. doi: 10.1519/JSC.0000000000001666. PMID 28640771
- [Background] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160